CLINICAL TRIAL: NCT06008054
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of SI-B003 Monotherapy, BL-B01D1+SI-B003 Combination Therapy and BL-B01D1+PD-1 Monoclonal Antibody in Patients With Locally Advanced or Metastatic Esophageal Cancer, Gastric Cancer, Colorectal Cancer and Other Gastrointestinal Tumors
Brief Title: A Study of SI-B003, BL-B01D1+SI-B003 and BL-B01D1+PD-1 Monoclonal Antibody in Patients With Locally Advanced or Metastatic Esophageal Cancer, Gastric Cancer, Colorectal Cancer and Other Gastrointestinal Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Collaborators: Baili-Bio (Chengdu) Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-SI-B003-201-05
Record Dates: First submitted 2023-08-16; First posted 2023-08-23 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Cancer; Gastric Cancer; Colorectal Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Colorectal Neoplasms | interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SI-B003, BL-B01D1+SI-B003 and BL-B01D1+PD-1 Monoclonal Antibody (Experimental): Participants received SI-B003, BL-B01D1+SI-B003 and BL-B01D1+PD-1 Monoclonal Antibody in the first cycle (3 weeks). Participants who had a clinical benefit could receive additional cycles of additional treatment. Administration will be discontinued because of disease progression or intolerable toxicity or for other reasons.
  Interventions: Drug: SI-B003; Drug: BL-B01D1; Drug: PD-1 Monoclonal Antibody

INTERVENTIONS:
Drug: SI-B003 — Administered by intravenous infusion every 3 weeks (Q3W).
Drug: BL-B01D1 — Administered by intravenous infusion for a cycle of 3 weeks.
  Other Names: iza-bren; izalontamab brengitecan; BMS-986507
Drug: PD-1 Monoclonal Antibody — Administration by intravenous infusion for a cycle of 3 weeks.

SUMMARY:
This phase II study is a clinical study to explore the efficacy and safety of SI-B003 Monotherapy, BL-B01D1+SI-B003 Combination Therapy and BL-B01D1+PD-1 Monoclonal Antibody in patients with locally advanced or metastatic esophageal cancer, gastric cancer, colorectal cancer and other gastrointestinal tumors.

DETAILED DESCRIPTION:
To explore the efficacy, safety and tolerability of SI-B003 Monotherapy, BL-B01D1+SI-B003 Combination Therapy and BL-B01D1+PD-1 Monoclonal Antibody in patients with locally advanced or metastatic esophageal cancer, gastric cancer, colorectal cancer and other gastrointestinal tumors, and to further explore the optimal dose and combination way.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form voluntarily and follow the protocol requirements;
2. Gender is not limited;
3. Age: ≥18 years old and ≤75 years old;
4. Expected survival time ≥3 months;
5. Patients with locally advanced or metastatic esophageal cancer, gastric cancer, colorectal cancer and other gastrointestinal tumors;
6. Agreed to provide primary tumors or metastases 2 years archive of tumor tissue samples or fresh tissue samples;
7. At least one measurable lesion meeting the RECIST v1.1 definition was required;
8. ECOG 0 or 1;
9. The toxicity of previous antineoplastic therapy has returned to ≤ grade 1 as defined by NCI-CTCAE v5.0;
10. No severe cardiac dysfunction, left ventricular ejection fraction ≥50%;
11. No blood transfusion, no use of cell growth factors and/or platelet-raising drugs within 14 days before screening, and organ function levels must meet the criteria;
12. Blood coagulation function: international standardization ratio of 1.5 or less, and the part activated clotting time live enzymes ULN 1.5 or less;
13. Urinary protein ≤2+ or ≤1000mg/24h;
14. For premenopausal women with childbearing potential, a pregnancy test must be performed within 7 days before starting treatment, serum or urine must be negative for pregnancy, and must be non-lactating; All enrolled patients (male or female) were advised to use adequate barrier contraception throughout the treatment cycle and for 6 months after the end of treatment.

Exclusion Criteria:

1. Antitumor therapy such as chemotherapy or biological therapy was used within 4 weeks or 5 half-lives before the first dose in this study; Mitomycin and nitrosoureas were administered within 6 weeks before the first dose; Oral drugs such as fluorouracil;
2. Cohort using BL-B01D1, previously treated with an ADC drug with topoisomerase I inhibitor as toxin; Immunomodulatory drugs were administered within 2 weeks before the first dose in this study;
3. Systemic corticosteroids were required within 2 weeks before the first dose of the study;
4. Had received immunotherapy and developed grade ≥3 irAE or grade ≥2 immune-related myocarditis according to the CSCO guidelines;
5. History of severe heart disease;
6. QT prolongation, complete left bundle branch block, III degree atrioventricular block;
7. Active autoimmune and inflammatory diseases;
8. Other malignant tumors were diagnosed within 5 years before the first dose in this study;
9. Presence of: a) poorly controlled diabetes mellitus before starting study treatment; b) poorly controlled hypertension; c) history of hypertensive crisis or hypertensive encephalopathy;
10. Pulmonary disease defined as grade ≥3 according to CTCAE v5.0; The patient was diagnosed with grade ≥1 radiation pneumonitis according to the RTOG/EORTC definition. Patients with existing or a history of interstitial lung disease;
11. Unstable thrombotic events requiring therapeutic intervention within 6 months before screening; Infusion-related thrombosis was excluded;
12. Patients with unstable pericardial effusion, pleural effusion, ascites and other serous cavity effusion;
13. Patients with active central nervous system metastasis;
14. Patients with a history of allergy to recombinant humanized antibody or human-mouse chimeric antibody or to any ingredient of BL-B01D1 or SI-B003;
15. Prior organ transplantation or allogeneic hematopoietic stem cell transplantation (Allo-HSCT);
16. Human immunodeficiency virus antibody positive, active tuberculosis, active hepatitis B virus infection or hepatitis C virus infection;
17. Active infections requiring systemic therapy, such as severe pneumonia, bacteremia, sepsis, etc;
18. Enrolled in another clinical trial within 4 weeks before the first dose of this study;
19. Patients who received live vaccine within 4 weeks before the first dose;
20. Patients with a history of mental illness or drug abuse who are unable to cooperate with clinical trial requirements;
21. The investigator did not consider it appropriate to apply other criteria for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to approximately 24 months
  ORR is defined as the percentage of participants, who has a CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions). The percentage of participants who experiences a confirmed CR or PR is according to RECIST 1.1.
Recommended Phase II Dose (RP2D) | Up to approximately 24 months
  The RP2D is defined as the dose level chosen by the sponsor (in consultation with the investigators) for phase II study, based on safety, tolerability, efficacy, PK, and PD data collected during the dose escalation study .

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to approximately 24 months
  The PFS is defined as the time from the first dose of medication to disease progression or death, whichever occurred first.
Disease control rate (DCR) | Up to approximately 24 months
  The DCR is defined as the percentage of participants who has a CR, PR, or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease [PD: at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD]).
Duration of response (DOR) | Up to approximately 24 months
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Treatment-Emergent Adverse Event (TEAE) | Up to approximately 24 months
  TEAE is defined as any adverse and unexpected change in body structure, function, or chemistry or any exacerbation of an existing condition (i.e., any clinically significant adverse change in frequency and/or intensity) during treatment. The type, frequency, and severity of TEAE will be assessed during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China